CLINICAL TRIAL: NCT00909948
Title: Intentional Rejection of the Donor Graft Using Recipient Leukocyte Infusion(s) Following Nonmyeloablative Allogeneic Stem Cell Transplant
Acronym: RLI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Bimalangshu Dey, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 07-068; NCT00981760 (obsolete NCT alias)
Record Dates: First submitted 2009-05-27; First posted 2009-05-29 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Non Hodgkin's Lymphoma; Hodgkin Disease; Multiple Myeloma
Keywords: Related stem cell transplant,; TBI,; Mismatched stem cell transplant; Fludarabine; Non-myeloablative; Lymphoma; Multiple myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Lymphoma | interventions — fludarabine; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fludarabine (Active Comparator): The patients in this cohort will receive fludarabine 30 mg/m2/day on days -4 to -2 and 200 cGy TBI on day 0.
  Interventions: Other: Fludarabine and total body irradiation
- TBI only (Active Comparator): Patients will be given 200 centiGray (cGy) total body irradiation (TBI) in one fraction. TBI will be given on day 0, 4 to 6 hours prior to HCT.
  Interventions: Radiation: Total body irradiation

INTERVENTIONS:
Other: Fludarabine and total body irradiation — The patients in the second cohort will receive fludarabine 30 mg/m2/day on days -4 to -2 and 200 cGy TBI on day 0.
  Arms: Fludarabine
Radiation: Total body irradiation — Patients will receive 200 cGy TBI on day 0,4-6 hours prior to HCT.
  Arms: TBI only

SUMMARY:
The proposed study is based on our observation of paradoxical tumor regression after rejection of the donor graft in conjunction with the results of our murine experiments. We hypothesize that clinically meaningful responses can be achieved in patients with advanced malignancies with a transplant strategy using nonmyeloablative conditioning and related mismatched donor stem cell transplant where the intention will be to initially achieve mixed chimerism which will be followed by recipient lymphocyte infusion (RLI) in an attempt to deliberately reject the donor graft. This will lead to the development of novel transplant strategies for achieving antitumor effects without the risk of graft versus host disease (GVHD). This proposed protocol is a Pilot Study that will evaluate the safety of this outpatient transplant strategy, i.e., establishment of initial mixed chimerism followed by RLI for donor graft rejection, in patients with advanced lymphomas, and multiple myeloma.

In addition, because RLI have been reported to reverse ongoing GVHD, this approach might potentially reverse GVHD while achieving antitumor responses if this complication unexpectedly occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chemorefractory non-Hodgkin's or Hodgkin's lymphoma or multiple myeloma.

   Criteria for consideration of enrollment will include:
   1. primary refractory or refractory relapsed disease for which autologous HCT is unlikely to be beneficial;
   2. relapse after autologous HCT
   3. ineligibility for standard myeloablative or nonmyeloablative allo-HCT because of either lack of a donor or patient considerations
2. Non Hodgkin's lymphoma, or Hodgkin's lymphoma: primary refractory or refractory relapse
3. Multiple myeloma; primary refractory or refractory relapse
4. Patients with the above malignancies who have had a previous autologous or allogeneic bone marrow or stem cell transplant.
5. An estimated disease-free survival of less than one year.
6. Age 18 to age < 75 years
7. ECOG performance status of 0, 1, or 2.

Exclusion Criteria:

1. Patients whose life expectancy is limited by diseases other than their malignancy
2. Patients who have a 5/6 or better matched related donor or a 4/6 or better umbilical cord blood donor and who are medically eligible for conventional myeloablative or non-myeloablative transplant will be excluded
3. Cardiac disease: symptomatic congestive heart failure or RVG or echocardiogram determined LVEF ogf< 30%, active angina pectoris or uncontrolled hypertension
4. Pulmonary disease: severe chronic obstructive lung disease, or symptomatic restrictive lung disease, or corrected DLCO < 40% of predicted
5. Renal disease: serum creatinine > 3.0 mg/dl.
6. Hepatic disease: serum bilirubin > 3.0 mg/dl or alkaline phosphatase, SGOT or SGPT > 3 x ULN
7. Neurologic disease: symptomatic leukoencephalopathy, active CNS malignancy or other neuropsychiatric abnormalities believed to preclude transplantation (pervious CNS malignancy presently in CR is not an exclusion)
8. Uncontrolled infection.
9. Recipient leukocyte infusion (RLI) might involve the infusion of circulating tumor cells to the patients. To minimize this risk patients who have evidence of circulating tumor cells by light microscopy and flow cytometry will be excluded
10. Patients with acute leukemia will be excluded because they will likely have much greater circulating tumor burden, which would increase the risk of infusion of clonal tumor cells

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To determine the safety at ≤100 days of a non myeloablative mismatched related HCT when followed by recipient leukocyte infusion to induce deliberate rejection of the donor graft. | 100 days post transplant

SECONDARY OUTCOMES:
To evaluate the incidence of acute and chronic GVHD | Up to 2 years post transplant
To evaluate the incidence of loss of donor grafts | Up to 2 years post transplant
To evaluate progression-free and overall survival | Up to 2 years post transplant
To evaluate antitumor responses following this transplant strategy | Up to 2 years post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Bimalangshu R Dey, MD, PhD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Bortin MM, Rimm AA, Saltzstein EC. Graft versus leukemia: quantification of adoptive immunotherapy in murine leukemia. Science. 1973 Feb 23;179(4075):811-3. doi: 10.1126/science.179.4075.811. PMID 4405359
- [Background] Hill GR, Krenger W, Ferrara JL. The role of cytokines in acute graft-versus-host disease. Cytokines Cell Mol Ther. 1997 Dec;3(4):257-66. PMID 9740354
- [Background] Dey BR, McAfee S, Colby C, Sackstein R, Saidman S, Tarbell N, Sachs DH, Sykes M, Spitzer TR. Impact of prophylactic donor leukocyte infusions on mixed chimerism, graft-versus-host disease, and antitumor response in patients with advanced hematologic malignancies treated with nonmyeloablative conditioning and allogeneic bone marrow transplantation. Biol Blood Marrow Transplant. 2003 May;9(5):320-9. doi: 10.1016/s1083-8791(03)00077-6. PMID 12766882
- [Background] Sykes M, Romick ML, Sachs DH. Interleukin 2 prevents graft-versus-host disease while preserving the graft-versus-leukemia effect of allogeneic T cells. Proc Natl Acad Sci U S A. 1990 Aug;87(15):5633-7. doi: 10.1073/pnas.87.15.5633. PMID 2377601
- [Background] Mapara MY, Kim YM, Wang SP, Bronson R, Sachs DH, Sykes M. Donor lymphocyte infusions mediate superior graft-versus-leukemia effects in mixed compared to fully allogeneic chimeras: a critical role for host antigen-presenting cells. Blood. 2002 Sep 1;100(5):1903-9. doi: 10.1182/blood-2002-01-0023. PMID 12176915
- [Background] Kraus AB, Shaffer J, Toh HC, Preffer F, Dombkowski D, Saidman S, Colby C, George R, McAfee S, Sackstein R, Dey B, Spitzer TR, Sykes M. Early host CD8 T-cell recovery and sensitized anti-donor interleukin-2-producing and cytotoxic T-cell responses associated with marrow graft rejection following nonmyeloablative allogeneic bone marrow transplantation. Exp Hematol. 2003 Jul;31(7):609-21. doi: 10.1016/s0301-472x(03)00082-1. PMID 12842706
- [Background] Spitzer TR, McAfee S, Sackstein R, Colby C, Toh HC, Multani P, Saidman S, Weyouth DW, Preffer F, Poliquin C, Foley A, Cox B, Andrews D, Sachs DH, Sykes M. Intentional induction of mixed chimerism and achievement of antitumor responses after nonmyeloablative conditioning therapy and HLA-matched donor bone marrow transplantation for refractory hematologic malignancies. Biol Blood Marrow Transplant. 2000;6(3A):309-20. doi: 10.1016/s1083-8791(00)70056-5. PMID 10905768
- [Background] Rubio MT, Kim YM, Sachs T, Mapara M, Zhao G, Sykes M. Antitumor effect of donor marrow graft rejection induced by recipient leukocyte infusions in mixed chimeras prepared with nonmyeloablative conditioning: critical role for recipient-derived IFN-gamma. Blood. 2003 Sep 15;102(6):2300-7. doi: 10.1182/blood-2002-12-3949. Epub 2003 Jun 5. PMID 12791660
- [Background] Ballen KK, Becker PS, Emmons RV, Fitzgerald TJ, Hsieh CC, Liu Q, Heyes C, Clark Y, Levy W, Lambert JF, Chiafari F, Szymanski I, Rososhansky S, Popovsky MA, Stewart FM, Quesenberry PJ. Low-dose total body irradiation followed by allogeneic lymphocyte infusion may induce remission in patients with refractory hematologic malignancy. Blood. 2002 Jul 15;100(2):442-50. doi: 10.1182/blood.v100.2.442. PMID 12091334
- [Background] Colby C, Sykes M, Sachs DH, Spitzer TR. Cellular modulation of acute graft-vs.-host disease. Biol Blood Marrow Transplant. 1997 Dec;3(6):287-93. PMID 9502295